CLINICAL TRIAL: NCT02176083
Title: Intervening on Reproductive Health in Young Breast Cancer Survivors
Brief Title: Reproductive Health Survivorship Care Plan Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Hui-Chun Irene Su, Assistant Professor of Reproductive Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCP-1
Record Dates: First submitted 2014-06-20; First posted 2014-06-26 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer; Hot Flashes; Vaginal Dryness; Estrogen Deprivation Symptoms
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Text message management prompts: YBCS will receive text message prompts on how to manage hot flashes and vaginal dryness
  Interventions: Behavioral: Text message management prompts
- Control (No Intervention): Control YBCS will not receive text message prompts on managing hot flashes and vaginal dryness

INTERVENTIONS:
Behavioral: Text message management prompts
  Arms: Intervention

SUMMARY:
Most young breast cancer patients undergo chemotherapy and/or endocrine therapy, treatments that impair ovarian function and result in significant reproductive health late effects. These late effects include symptoms of estrogen deprivation (e.g., hot flashes and vaginal dryness), which are distressing in young breast cancer survivors (YBCS). The goal of this pilot study is to test the feasibility of a 4-week text message based intervention on hot flashes and vaginal dryness in YBCS. YBCS will be randomized in a 1:1 ratio to the intervention (text messages on hot flash and vaginal dryness management) and control arms. All participants will be prompted to provide daily hot flash frequency and severity via text messaging. The primary hypothesis is YBCS will have high rates of daily hot flash reporting via text messaging. Secondarily, we will compare changes in hot flash frequency, hot flash severity and vagina dryness between the intervention and control arms.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer
* Female
* Completed primary breast cancer treatment
* Age <=45

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-03-20; Primary Completion 2014-08-31 (Actual); Study Completion 2015-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Su, MD MSCE, Principal Investigator — UC San Diego
Locations (2):
- United States (2):
  - UC San Diego, La Jolla, California
  - UCSD Moores Cancer Center, La Jolla, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Text message management prompts: YBCS will receive text message prompts on how to manage hot flashes and vaginal dryness
  Text message management prompts
Period: Overall Study
Arm/Group | Intervention | Control
Started | 11 | 27
Completed | 11 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 11 | 27 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 27 | 38
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 27 | 38
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 27 | 38

OUTCOME MEASURES:

1. Primary Outcome: Hot Flash Frequency
Description: Median number of daily hot flashes over 4th week of study
Time Frame: 1 week
Measure: Median (Inter-Quartile Range); unit: daily hot flashes
Arm/Group | Intervention | Control
Number analyzed (Participants) | 11 | 27
daily hot flashes | 2.2 [1.2 to 3.6] | 1.4 [0.7 to 2.3]

ADVERSE EVENTS:
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/27
Other Adverse Events (participants affected / at risk) | 0/11 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No